CLINICAL TRIAL: NCT04516915
Title: Prospective, Randomized, Parallel-Group, Open-Label Study to Evaluate the Efficacy and Safety of IMU-838, in Combination With Oseltamivir, in Adults With COVID-19
Brief Title: IMU-838 and Oseltamivir in the Treatment of COVID-19
Acronym: IONIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Immunic AG (Industry); University of Warwick (Other); MODEPHARMA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA486120
Record Dates: First submitted 2020-08-10; First posted 2020-08-18 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Covid 19
MeSH Terms: conditions — COVID-19 | interventions — Oseltamivir

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Parallel-Group, Open-Label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMU-838 + Oseltamivir (Experimental): Loading dose of IMU-838 followed by 22.5mg BID plus Oseltamivir (75mg BID) for 14 days
  Interventions: Drug: IMU-838; Drug: Oseltamivir
- Oseltamivir (Active Comparator): Oseltamivir (75mg BID) for 14 days
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: IMU-838 — IMU-838 twice daily at 22.5mg doses for 14 days
  Other Names: Intervention Arm
  Arms: IMU-838 + Oseltamivir
Drug: Oseltamivir — Oseltamivir twice daily at 75mg doses for 14 days
  Other Names: Control arm

SUMMARY:
To evaluate whether time-to-improvement is significantly better in IMU-838 plus Oseltamivir (IONIC Intervention) and standard care vs. Oseltamivir and standard care in adult subjects with coronavirus disease (COVID-19)

DETAILED DESCRIPTION:
The IONIC Protocol describes an overarching trial design to provide reliable evidence on the efficacy of IMU-838 (vidofludimus calcium) when delivered in combination with an antiviral therapy (Oseltamivir) [IONIC Intervention] for confirmed or suspected COVID-19 infection in adult patients receiving usual standard of care.

At present, there are no known treatments for COVID-19. Whilst, the anticipated scale of the epidemic is such that hospitals, and particularly intensive care facilities, may be massively overstretched. As described by a few models of pandemic spread, up to 50% of the adult population may fall sick over a period of 8-12 weeks, of whom around 10% may require hospitalisation. This figure could imply nearly 2 million hospital admissions. Considering this scenario, therapies which may only have a moderate impact on survival or on hospital resources could be worthwhile.

Critically, the present trial design has been developed with consideration of the front-line hospital staff working within an overstretched care system in these unprecedented times. To minimise their burden the protocol is deliberately flexible so that it is suitable for a wide range of settings, allowing:

* a broad range of patients to be enrolled (patient pathway, disease stage or mode of diagnosis)
* Additional sub-studies may be added to provide more detailed information on side effects or sub-categorisation of patient types but these are not the primary objective and are not required for participation.
* To be able to include more sites: the investigators will initiate the trial as a single centre (UHCW) and more sites invited to participate according to the emerging evidence
* The investigator have included 'Exploratory and Secondary objectives' in the protocol however, in consideration of the circumstances the research activities will emulate investigations performed as per standard care/routines care to minimise any burden on the delivery teams.

This is a Phase 2b, randomised, parallel-group, open-label study to assess the efficacy and safety of an oral dose of IMU-838 (22.5 mg twice daily [45 mg/day]) plus Oseltamivir (75mg twice daily [150mg/day]) (IONIC Intervetion) or Oseltamivir alone (75mg twice daily) in hospitalised patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or non-pregnant female patients at least 18 years old 2. Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 infection, either:

  * Confirmed cases: prospective participants who test positive to a validated specific SARS-CoV-2 nucleic acid test or has the virus identified by electron microscopy or viral culture, as per local trust policy ≤ 7 days before randomisation.
  * Probable/Suspected case: prospective participants who may have been in contact with a confirmed case of COVID-19, AND have mild to severe COVID-19 clinical symptoms AND radio-graphic evidence* of pulmonary infiltrates consistent with COVID-19 disease 3. Moderate to severe COVID-19 requiring hospitalisation defined as: a) Clinical status category 3-5 (inclusive) on the 7-point clinical status category scale as proposed by the World Health Organisation (WHO) master protocol: I. Category 3: hospitalized, no oxygen therapy II. Category 4: hospitalized, oxygen by mask or nasal prongs III. Category 5: hospitalized, non-invasive ventilation or high-flow oxygen *where routinely available, no tests will be requested for research purpose

Exclusion Criteria

Therapy Exclusion Criteria:

Use of the following concomitant medications is prohibited at Screening Visit and throughout the duration of the trial:

1. Use of Oseltamivir for more than 48 hrs prior to the first treatment dose
2. Use of antiviral drugs (e.g. nucleoside analogue reverse-transcriptase inhibitors, protease inhibitors, etc.)
3. History of long-term or concurrent use of mycophenolate mofetil, methotrexate exceeding 17.5 mg weekly
4. Chloroquine or hydroxychloroquine
5. Any medication known to significantly increase urinary elimination of uric acid, in particular lesinurad as well as uricosuric drugs such as probenecid
6. Treatments for any malignancy, in particular irinotecan, paclitaxel, tretinoin, bosutinib, sorafinib, enasidenib, erlotinib, regorafenib, pazopanib and nilotinib
7. Any drug significantly restricting water diuresis, in particular vasopressin and vasopressin analogues
8. Use of rosuvastatin at daily doses higher than 10 mg

Medical History of Concomitant Disease Exclusion Criteria

* Allergic or hypersensitivity to the IMU-838, Oseltamivir, or any of the ingredients
* Pregnant or breastfeeding or with intention to become pregnant during the study
* Participants who cannot take trial medication orally at presentation
* Undergoing active chemotherapy or radiotherapy.
* If the attending clinician believes that there is a specific contra-indication to the IONIC intervention.
* Patient has a medical or concomitant disease history preventing them from participating
* Critical patients whose expected survival time < 48-72 hours
* Evidence of pancytopenia or immunosuppression
* Any contraindication to Oseltamivir or standard of care

Presence of the following laboratory values at Screening Exclusion Criteria

* Platelet count <100,000/mm³ (<100 x 109/L)
* Total bilirubin > 2 x ULN or ALT or GGT > 5 x ULN
* Elevated indirect (unconjugated) bilirubin >1.2 x ULN (i.e. >1.1 mg/dL)
* Serum uric acid levels at Screening Visit >1.2 x ULN (for women >6.8 mg/dL, for men >8.4 mg/dL)
* Renal impairment defined as estimated glomerular filtration rate ≤45 mL/min/1.73m²
* Decompensated liver cirrhosis (Child-Pugh score B and C)
* History or presence of serious or acute heart disease such as uncontrolled cardiac dysrhythmia or arrhythmia, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure (New York Heart Association [NYHA] class 3 or 4)
* Cardiac disease resulting in marked limitation of physical activity. Patients are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain. NYHA class 4: Cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
* History or presence of any major medical or psychiatric illness (such as severe depression, psychosis, bipolar disorder), history of suicide attempt, or current suicidal ideation, if any of those conditions in the opinion of the investigator could create undue risk to the patient or could affect adherence with the trial protocol

COVID-19 related exclusion criteria

• Participation in any other interventional clinical trial for an experimental treatment for COVID-19

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
To evaluate whether time-to-improvement is significantly better in IMU-838 plus Oseltamivir (IONIC Intervention) vs. Oseltamivir alone in adult subjects with COVID-19 | 14 days
  Time-to-clinical improvement; defined as the time from randomisation to a 2-point improvement on the world health organizations 9-point ordinal scale (ranging from 0-8; 0 being no evidence of clinical infection and 8 being death), discharge from hospital, or death (whichever occurs first)

SECONDARY OUTCOMES:
To evaluate safety (number of adverse events) and tolerability (laboratory abnormalities) of IMU 838 + Oseltamivir vs. Oseltamivir alone in adult subjects with COVID-19. | 28 days
  Incidence of Adverse events (AEs) and serious adverse events (SAEs), including COVID-19 worsening and incidence of laboratory abnormalities (defined as a 1.5x increase in liver function test results (total protein, albumin, bilirubin, alkaline phosphotase and ALT) from screening).
To determine the effects of IONIC Intervention on improvement of at least two points in clinical status scale (from 0 to 8; with 8 being no evidence of clinical infection and 8 being death) | 28 days
  Proportion of patients with two-point change on WHO ordinal scale at Day 7 and 28
To assess the effects of IONIC Intervention vs. Oseltamivir on the need for invasive ventilation, renal replacement therapy or ECMO | 14 days
  Proportion of patients free of invasive ventilation, renal replacement therapy or ECMO at Day 7 and 14
To assess the effects of IONIC Intervention vs. Oseltamivir on the length of hospital and intensive care unit (ICU) stay | 28 days
  To assess the effects of IONIC Intervention vs. Oseltamivir on the length of hospital and intensive care unit (ICU) stay
To assess the effects of IONIC Intervention vs. Oseltamivir on the time from treatment initiation to death | 28 days
  Mortality at day 28 and time from treatment initiation to death

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Coventry and Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma K, Berry L, Vryonis E, Ali A, Lara B, Noufaily A, Parsons N, Bradley C, Haley B, Tabuso M, Arasaradnam RP. Prospective, randomised, parallel-group, open-label study to evaluate the effectiveness and safety of IMU-838, in combination with oseltamivir, in adults with COVID-19: the IONIC trial protocol. BMJ Open. 2022 Nov 17;12(11):e055205. doi: 10.1136/bmjopen-2021-055205. PMID 36396307